CLINICAL TRIAL: NCT06087146
Title: Sauerkraut Supplementation in Athletes for Gut Microbiome Optimization: Case Series and Literature Review (Project KOMS)
Brief Title: Modulation of the Gut Microbiota of Professional Athletes With Sauerkraut Supplementation
Acronym: KOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Gut Microbiome Center (Centar za crijevni mikrobiom) (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KOMS77
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Microbiome
Keywords: Microbiota; Sports; Athletes; Nutrition Surveys; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes supplemented with sauerkraut (Experimental): 10 professional athletes (9 male) who will during 10 days consume approximately 250 g of sauerkraut (Brassica oleracea v. capitata) daily.
  Interventions: Other: Sauerkraut (Brassica oleracea v. capitata)

INTERVENTIONS:
Other: Sauerkraut (Brassica oleracea v. capitata) — The research material is a donation from the company Eko Bio Zrnje, Vrbovec, Croatia. It's grated pickle cabbage produced by fermentation in a saline solution (NaCl) in which the fermentation was stopped by pasteurization and was packed in glass 500g jars. The nutritional and microbiological composition was tested by the laboratories of the Faculty of Food and Biotechnology, as well as by the cultural laboratory approach confirmed the presence of bacteria that produce lactic acid (4.82·103 (±2.31) CFU/mL)

SUMMARY:
Literature on the topic of athlete gut microbiota is scarce, and even more on the topic of its modulation.

To address these issues a prospective cohort study was conceived. The cohort included young, male generally healthy professional athletes. The cohort will first be exposed to a course of sauerkraut supplementation as a synbiotic. Then the cohort will be observed without any intention for gut microbiota modulation. Before and after each study phase a gut microbiota analysis will be performed for its parameters. The aim of this study is to assess whether the intervention leads to significant changes in the gut microbiota parameters in all subjects and if yes what the signal of the intervention was, meaning whether the changes were consistent among all subjects regarding the analyzed parameter and its direction of effect. The results will be compared with data from earlier research on gut microbiota modulation in professional athletes with soluble fiber as prebiotics and a placebo. The study will provide valuable data on the athlete gut microbiota and its potential modulation.

DETAILED DESCRIPTION:
Material, participants, methodology and research plan The subject of the research will be interventions with sauerkraut to modulate the intestinal microbiota as a synbiotic as a substance whose effect has been established in previous scientific research on humans, and which, due to the low incidence of side effects, have been assessed as generally safe. The intervention will refer to the use of sauerkraut. During 10 days, the subjects will consume approximately 250 g of sauerkraut (Brassica oleracea v. capitata) daily. The research material is a donation from the company Eko Bio Zrnje, Vrbovec, Croatia. It's grated pickle cabbage produced by fermentation in a saline solution (NaCl) in which the fermentation was stopped by pasteurization and was packed in glass 500g jars. The nutritional and microbiological composition was tested by the laboratories of the Faculty of Food and Biotechnology, as well as by the cultural laboratory approach confirmed the presence of bacteria that produce lactic acid (4.82·103 (±2.31) colony forming unit/mL) with potential probiotic due to which this product can be considered a synbiotic. Additionally, sauerkraut was analyzed using 16s ribosomal ribonucleic acid natural guide star next-generation sequencing nonconvulsive generalized status epilepticus normal goat serum methods on the presence of genetic material of bacteria within it. With regard to pasteurization, sauerkraut will not be necessary transport and store according to the cold chain principle. The results of the intervention regarding the modulation of the intestinal microbiota will be compared with those from the previous research in which the subject is research was the modulation of intestinal microbiota by soluble fiber NUTRIOSE in professional athletes. NUTRIOSE are resistant maltodextrin, i.e. non-viscous soluble fibers obtained from wheat and corn (Roquette Freres, Lestrem, France) with proven prebiotic action.

respondents For the purposes of the research, a cohort will be formed with a minimum of nine respondents - professional athletes. The sample of respondents was determined technical, logistical and financial conditions of the research, and is based on the fact that the comparison with cohorts of 9 subjects from a previous study (NCT05726435) who were exposed to the intervention with prebiotics and controlled by placebo with the aim modulation of the intestinal microbiota of professional athletes. The recruitment of respondents will be carried out in cooperation with research partners (HOO) and from the researcher's social environment using an online questionnaire.

Methodology

Work methods: dietetic methods, anthropometric methods and collection and analysis of venous blood and stool samples. The sample of variables consists of: a sample of feces for sequencing the intestinal microbiota, a sample of venous blood for laboratory processing, measures for the assessment of morphological characteristics (body height, body mass, percentage of fat tissue and muscle tissue calculated using the analyzer for body composition - TANITA bioimpedance). Dietetic methods will be used to control the intake of all nutrients before and during the intervention as well as during the follow-up phase. From the method will be a food diary (seven-day and ten-day). All collected dietary data will be processed through Capnutr atlas of foodstuffs and ready meals from the Balkan region (Glibetić et al., 2018).

Research plan The research was designed as a prospective cohort study. The research will be conducted in compliance with the regulations of the Declaration of Helsinki and in accordance with the approval of the Ethics Committee of the Faculty of Medicine of the University of Zagreb dated 27.3.2023. Research will to be carried out in two phases: in the first phase, the subjects will be supplemented with sauerkraut for ten days, and in the second phase of one month will be monitored for intestinal microbiota without attempting to modulate the intestinal microbiota ("wash-out"). In cooperation with HOO and academic and business partners, professional athletes will be invited to fill out the virtual form "Athletes and intestinal microbiome", that is, a questionnaire about athletes' knowledge about the intestinal microbiome. Data processing will identify potential candidates for Research. Candidates will be contacted by phone, informed about the research and evaluated in a short conversation regarding the criteria on and off. Candidates who meet the criteria will be included in the cohort. After the establishment of the cohort, logistical arrangements will be made and study plan plan. The study will be divided into three phases: before, during and after the intervention. First, the subjects will be informed about the study plan (time, number of visits, logistics) for which informed consent was obtained. In the pre-intervention phase, there will be a meeting in which more once explain the plan and course of the study, define the deadlines and distribute the equipment for taking the sample and send the provided forms (Excel, Microsoft Office, USA). In the continuation of the first phase, the respondents will record daily food intake, duration and intensity of physical activity as well as sleep time. Likewise, questionnaires on the question of the quality of diet (DQQ), a questionnaire on knowledge about nutrition and chronotype questionnaire. The day before the start of the intervention, the subjects will provide a stool and blood sample, and then fill out the acceptable daily intake. During the intervention respondents are in continuous communication with the team of researchers. In a specially provided form, they record adherence to the intervention (data i time of intake of cabbage, for example) and possible side effects (changes in the stool, flatulence, wind) as well as the type of stool according to the Bristol scale. During intervention subjects continue to keep a diet, exercise and sleep diary. After the intervention, they give a blood sample again and a sample of the first one chairs after the intervention, according to the same principle as before the intervention. Likewise, the respondents will fill out the ADI again. In the second phase research subjects remain in communication with the researchers, and two months after the last stool sample is taken again a stool sample from the subject and the analysis of the intestinal microbiota is performed again. During data processing, the results of this research will be compared with the results of the previous research, which is different from this one research used prebiotics and not synbiotic in the intervention. Previous research registered in the ClinicalTrials.gov registry under no NCT05726435 was designed as a randomized placebo-controlled intervention study. The respondents, professional athletes, were during the 4 weeks, one group received either prebiotics, NUTRIOSE fibers, or a placebo in the amount of 20g divided into two doses of 10g each. Analysis intestinal microbiota were performed on several occasions during the described intervention. The results of this research will be compared specifically with the results of the intestinal microbiota analysis at two time points: after 2 weeks of the intervention and 8 weeks from the start of the intervention, when the subjects were 4 weeks without prebiotics or placebo after the intervention itself.

Data processing methods:

Differences between categorical variables will be tested using the chi-square test. Differences between non-categorical variables will be examined, depending on distribution and number of groups, paired t-test as well as Kruskal-Wallis and Mann-Whitney U test and then Bonferoni test for post hoc analysis.

In order to examine possible correlations, the calculation of Pearson correlation coefficients between parameters of nutritional status will be used, body composition and diet. The questionnaires will be validated by calculating the Cronbach alpha coefficient for each of their items and through an exploratory one factor analysis, and internal consistency will be determined by calculating Pearson's correlation coefficients between individual items questionnaire. The relative shares of individual taxonomic categories will be used to calculate the Shannon-Wiener diversity index in order to compared the diversity between the group of samples before and after the intervention. Cluster analysis will be performed using the BioNumerics program (Applied Maths, Belgium) based on Haemophilus haemolyticus restriction endonuclease I and MSPi T-restriction fragment length polymorphism patterns. P values below 0.05 will be considered statistically significant. For statistical data processing will be carried out using the SPSS 19.0 program (IBM, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* regularly engaging in professional sports activities

  1. categorized athlete by HOO
  2. playing sports as a source of income (bodybuilding)
* older than 18 years old
* general general state of health
* written understanding of the English language

Exclusion Criteria:

* use of antibiotics for a period of at least six months before participating in the study application of nutritional supplements with the potential to modulate intestinal microbiota (probiotics, prebiotics, postbiotics) in the period from
* at least six months before participating in the study
* chronic drug therapy
* intolerance of one of the interventions (sauerkraut, fasting, probiotics and their additives)
* chronic medical therapy (except for vitamins, thyroid hormones and antihistamines)
* kidney function disorder
* liver function disorder
* history of digestive problems at the time before the study (diarrhea, dyspepsia, constipation)
* hormonal disorder (except hypothyroidism)
* psychological or mental disorder
* involvement in other research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Current | one month
  -short term gut microbiota change-
  The impact of sauerkraut on gut microbiome shall assessed through monitoring of relative taxonomic abundance of bacteria that compose gut microbiota from samples taken day before the intervention and immediately after the intervention.
  The composition of the intestinal microbiota will be determined by sequencing the 16s rRNA bacteria in the stool sample. Subjects take a sample with a sterile cotton swab by wiping stool with toilet paper in their home on a given day research. The sample is stored in a tube with a buffer liquid so that the sample can be stored and transported at room temperature temperature. The test sample is transported by air to the laboratory of Biomes NGS Gesellschaft mit beschränkter Haftung, Wildau, Germany. The laboratory performs independently

SECONDARY OUTCOMES:
Future | three months
  -long term gut microbiota change-
  After two months from the last stool sample,the respondents takes again a stool sample from the subject, and the analysis of the intestinal microbiota is performed again as described in the previous section.
  -comparison with similar study-
  During data processing, the results of this research will be compared with the results of the previous research, which is different from this one research used prebiotics and not synbiotics in the intervention. Previous research registered in the ClinicalTrials.gov registry under no NCT05726435 was designed as a randomized placebo-controlled intervention study. The respondents, professional athletes, were during the 4 weeks, one group received either prebiotics, NUTRIOSE fibers, or a placebo in the amount of 20g divided into two doses of 10g each.

CONTACTS AND LOCATIONS:
Locations (1):
- Gut Microbiome Center, Zagreb, Croatia

REFERENCES:
- [Result] Nichols AW. Probiotics and athletic performance: a systematic review. Curr Sports Med Rep. 2007 Jul;6(4):269-73. PMID 17618005
- [Result] Jager R, Mohr AE, Carpenter KC, Kerksick CM, Purpura M, Moussa A, Townsend JR, Lamprecht M, West NP, Black K, Gleeson M, Pyne DB, Wells SD, Arent SM, Smith-Ryan AE, Kreider RB, Campbell BI, Bannock L, Scheiman J, Wissent CJ, Pane M, Kalman DS, Pugh JN, Ter Haar JA, Antonio J. International Society of Sports Nutrition Position Stand: Probiotics. J Int Soc Sports Nutr. 2019 Dec 21;16(1):62. doi: 10.1186/s12970-019-0329-0. PMID 31864419
- [Result] Toohey JC, Townsend JR, Johnson SB, Toy AM, Vantrease WC, Bender D, Crimi CC, Stowers KL, Ruiz MD, VanDusseldorp TA, Feito Y, Mangine GT. Effects of Probiotic (Bacillus subtilis) Supplementation During Offseason Resistance Training in Female Division I Athletes. J Strength Cond Res. 2020 Nov;34(11):3173-3181. doi: 10.1519/JSC.0000000000002675. PMID 33105368
- [Result] Mohr AE, Pugh J, O'Sullivan O, Black K, Townsend JR, Pyne DB, Wardenaar FC, West NP, Whisner CM, McFarland LV. Best Practices for Probiotic Research in Athletic and Physically Active Populations: Guidance for Future Randomized Controlled Trials. Front Nutr. 2022 Mar 8;9:809983. doi: 10.3389/fnut.2022.809983. eCollection 2022. PMID 35350412
- [Result] Marco ML, Hutkins R, Hill C, Fulgoni VL, Cifelli CJ, Gahche J, Slavin JL, Merenstein D, Tancredi DJ, Sanders ME. A Classification System for Defining and Estimating Dietary Intake of Live Microbes in US Adults and Children. J Nutr. 2022 Jul 6;152(7):1729-1736. doi: 10.1093/jn/nxac074. PMID 35583208
- [Result] Dimidi E, Cox SR, Rossi M, Whelan K. Fermented Foods: Definitions and Characteristics, Impact on the Gut Microbiota and Effects on Gastrointestinal Health and Disease. Nutrients. 2019 Aug 5;11(8):1806. doi: 10.3390/nu11081806. PMID 31387262
- [Result] Touret T, Oliveira M, Semedo-Lemsaddek T. Putative probiotic lactic acid bacteria isolated from sauerkraut fermentations. PLoS One. 2018 Sep 7;13(9):e0203501. doi: 10.1371/journal.pone.0203501. eCollection 2018. PMID 30192827
- [Result] Costa MS, Toscano LT, Toscano LLT, Luna VR, Torres RA, Silva JA, Silva AS. Ergogenic potential of foods for performance and recovery: a new alternative in sports supplementation? A systematic review. Crit Rev Food Sci Nutr. 2022;62(6):1480-1501. doi: 10.1080/10408398.2020.1844137. Epub 2020 Nov 23. PMID 33226268
- [Result] Hughes RL, Holscher HD. Fueling Gut Microbes: A Review of the Interaction between Diet, Exercise, and the Gut Microbiota in Athletes. Adv Nutr. 2021 Dec 1;12(6):2190-2215. doi: 10.1093/advances/nmab077. PMID 34229348